CLINICAL TRIAL: NCT00537095
Title: A Randomized, Double Blind, Placebo-controlled Phase II, Multi-Centre Study to Assess the Efficacy and Safety of Vandetanib (ZD6474) in Patients With Locally Advanced or Metastatic Papillary or Follicular Thyroid Carcinoma Failing or Unsuitable for Radioiodine Therapy
Brief Title: Efficacy and Safety of Vandetanib (ZD6474) in Patients With Metastatic Papillary or Follicular Thyroid Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D4200C00079; 2007-001890-27 (EudraCT Number); LPS14940 (Other: Sanofi)
Record Dates: First submitted 2007-09-27; First posted 2007-09-28 (Estimated); Results first posted 2011-07-08 (Estimated); Last update posted 2024-04-19 (Actual); Status verified 2023-11

CONDITIONS: Thyroid Neoplasms
Keywords: follicular; papillary
MeSH Terms: conditions — Thyroid Neoplasms | interventions — vandetanib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- vandetanib (ZD6474) (Experimental): vandetanib (ZD6474) 300 mg per os once daily
  Interventions: Drug: Vandetanib
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Vandetanib — 300 mg oral once daily oral dose
  Other Names: SAR390530
  Arms: vandetanib (ZD6474)
Other: Placebo
  Arms: Placebo

SUMMARY:
This was a parallel group, randomized, double blind, placebo controlled, multicentre study designed to assess whether vandetanib (ZD6474) conferred an improvement in PFS as compared to placebo in participants with locally advanced or metastatic papillary or follicular thyroid carcinoma failing or unsuitable for radioiodine therapy. The trial was of a sufficient size so that if vandetanib (ZD6474) was truly active there was a high probability that it would demonstrate an effect sufficiently promising to warrant a follow-up assessment.

* Participants were seen weekly for the first 2 weeks, then again at Week 4, Week 8, and Week 12 after randomization, and every 12 weeks thereafter. Upon disease progression, all participants (both active and placebo) were unblinded and given the option to discontinue blinded study treatment and enter follow up and survival, or begin open label vandetanib (ZD6474) 300 mg treatment. All participants were followed to collect survival data until greater than or equal to (>=) 50% of participants had died. Participants who were taking vandetanib (ZD6474) at the time of study closure and wished to remain on therapy were allowed to continue for as long as the Investigator felt that they were obtaining clinical benefit, or until they were given another anti-cancer therapy. The safety data from all participants was assessed on an ongoing basis, including discontinuation and follow up.
* Radiologic evaluation using RECIST criteria was performed every 12 weeks (+/- 2 weeks). All medical images were centralized assessed at the site and centrally reviewed. Participants were evaluated until progression, and then followed up for survival, regardless of whether they continued randomized treatment, unless they withdrew consent. Post progression open-label vandetanib (ZD6474) were offered at the investigators discretion.
* All participants submitted a suitable archived tumor sample prior to randomization. In the event that a suitable archived sample was not available within 2 weeks prior to randomization, a fresh tumor sample was obtained in its place prior to randomization. If a participant underwent the fresh tumor biopsy procedure, this specimen would satisfy the first optional tumor biopsy submission should they consented to the exploratory part of the study.

ELIGIBILITY:
Inclusion Criteria:

* Previously confirmed histological diagnosis of locally advanced or metastatic papillary or follicular thyroid carcinoma, without anaplastic component. Tumor sample available for centralized exploratory analysis.
* Presence of one or more measurable lesions at least 1 cm in the longest diameter by spiral CT scan or 2 cm with conventional techniques.
* Progressive disease following RAI131 or patient unsuitable for RAI131 after surgery.
* Serum TSH <0.5 mU/L.

Exclusion Criteria:

* Major surgery within 4 weeks before randomization.
* Prior chemotherapy within the last 4 weeks prior to randomization.
* RAI131 therapy within 3 months in patients with radioiodine uptake.
* Radiation therapy within the last 4 weeks prior to randomization (with the exception of palliative radiotherapy).
* Serum bilirubin >1.5*the upper limit of reference range (ULRR).
* Creatinine clearance < 30 ml/min (calculated by Cockcroft-Gault formula).
* Alanine aminotransferase (ALT), aspartate aminotransferase (AST), or alkaline phosphatase (ALP) greater than 2.5*ULRR, or greater than 5.0*ULRR if judged by the investigator to be related to liver metastases.
* Clinically significant cardiovascular event (eg myocardial infarction), superior vena cava [SVC] syndrome, New York Heart Association [NYHA] classification of heart failure >II within 3 months before entry, or presence of cardiac disease that in the opinion of the Investigator increases the risk of ventricular arrhythmia.
* History of arrhythmia (multifocal premature ventricular contractions [PVCs], bigeminy, trigeminy, ventricular tachycardia or uncontrolled atrial fibrillation), which is symptomatic or requires treatment (CTCAE grade 3), , or asymptomatic sustained ventricular tachycardia. Participants with atrial fibrillation controlled by medication are permitted.
* Congenital long QT syndrome or 1st degree relative with unexplained sudden death under 40 years of age.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2007-09-28 (Actual); Primary Completion 2009-12-02 (Actual); Study Completion 2021-11-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Chair — Sanofi
Locations (15):
- Research Site, Brussels, Belgium
- Research Site, Odense, Denmark
- France (7):
  - Research Site, Angers
  - Research Site, Bordeaux
  - Research Site, Caen
  - Research Site, Lyon
  - Research Site, Marseille
  - Research Site, Paris
  - Research Site, Villejuif
- Research Site, Oslo, Norway
- Spain (2):
  - Research Site, L'Hospitalet de Llobregat
  - Research Site, Madrid
- Sweden (2):
  - Research Site, Lund
  - Research Site, Stockholm
- Research Site, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Leboulleux S, Bastholt L, Krause T, de la Fouchardiere C, Tennvall J, Awada A, Gomez JM, Bonichon F, Leenhardt L, Soufflet C, Licour M, Schlumberger MJ. Vandetanib in locally advanced or metastatic differentiated thyroid cancer: a randomised, double-blind, phase 2 trial. Lancet Oncol. 2012 Sep;13(9):897-905. doi: 10.1016/S1470-2045(12)70335-2. Epub 2012 Aug 14. PMID 22898678
- See also: Related Info — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_6111&studyid=353&filename=CSR-D4200C00079.pdf
- See also: CSR-D4200C00079.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_6111&studyid=353&filename=CSR-D4200C00079.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 164 participants were enrolled in the study, out of which only 145 participants were randomized into 2 arms to receive vandetanib 300 mg once daily oral dose or placebo. Participants were randomized by 16 active centers in 7 European countries from September 28th, 2007 to October 16th, 2008.
Pre-assignment Details: The main reason for non-randomization was non-respect of eligibility criteria.
Groups:
- ZD6474/ ZD6474: Participants received vandetanib (ZD6474) 300 mg orally once daily, until disease progression or until 12 months of stable disease during randomized treatment period, or until the end of the trial whichever comes first. Participants still receiving vandetanib (ZD6474) treatment at the end of the trial were offered the opportunity to enter the open label phase and continue to receive vandetanib (ZD6474) treatment as long as they still benefitted of it per investigator judgment or until subsequent anti-cancer therapy.
- PLACEBO/ ZD6474: Participants received placebo matching to vandetanib (ZD6474) tablet orally once daily, until disease progression or until 12 months of stable disease during randomized treatment period, or until the end of the trial whichever occurred first. Participants who experienced disease progression during the randomized phase were offered to enter the open-label phase and receive vandetanib (ZD6474) if, as long as they benefitted of it or until subsequent anti-cancer therapy.
Period: Randomized Treatment Period (433 Days)
Arm/Group | ZD6474/ ZD6474 | PLACEBO/ ZD6474
Started | 72 | 73
Safety Population | 73 (One participant in placebo arm received vandetanib (ZD6474) and was thus accounted in the vandetanib group for safety analysis.) | 72
Completed | 0 | 0
Not Completed | 72 | 73
Not completed — Adverse Event | 24 | 4
Not completed — Objective Disease Progression | 21 | 48
Not completed — Death | 3 | 1
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Subjective/ Clinic Progression or Lack of Efficacy | 1 | 2
Not completed — As per protocol (after 12 months of blinded treatment) | 21 | 16
Period: Open-label Period (590 Days)
Arm/Group | ZD6474/ ZD6474 | PLACEBO/ ZD6474
Started (Post completion of randomized treatment period, the participants were given the option to enter the open label period. In the open-label period, all participants received vandetanib (ZD6474).) | 28 | 59
Safety Population | 29 (One participant in placebo arm of randomized treatment period received vandetanib (ZD6474) and was thus accounted in the vandetanib group for the safety analysis.) | 58
Completed | 16 | 20
Not Completed | 12 | 39
Not completed — Adverse Event | 2 | 11
Not completed — Objective Disease Progression | 2 | 21
Not completed — Death | 2 | 2
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Subjective/ Clinic Progression or Lack of Efficacy | 5 | 3

BASELINE CHARACTERISTICS:
Population: Analysis was performed on intent to treat (ITT) population which included all randomized participants who received at least one dose of study treatment.
Groups:
- ZD6474: ZD6474, Vandetanib 300mg
- Total: Total of all reporting groups
Arm/Group | ZD6474 | PLACEBO | Total
Number analyzed (Participants) | 72 | 73 | 145
Age, Continuous [Mean (Standard Deviation); unit: year] | 62.8 (11.21) | 63.8 (11.59) | 63 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 34 | 67
  Male | 39 | 39 | 78

OUTCOME MEASURES:

1. Primary Outcome: Time to Tumor Progression
Description: modified RECIST V1.0 was used.
Time Frame: Time from date of randomization to date of the first documented tumor progression or date of death from any cause (within the 3 months) of tumor assessment
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | ZD6474 | PLACEBO
Number analyzed (Participants) | 72 | 73
days | 334 [232 to 421] | 176 [119 to 267]

2. Secondary Outcome: Disease Control Rate at 6 Months
Description: number of participants that achieved disease control 6 months after randomization. Best objective response of complete response + partial response + stable disease > 24 weeks according to RECIST criteria
Time Frame: 6 months after randomization
Measure: Number; unit: participants
Arm/Group | ZD6474 | PLACEBO
Number analyzed (Participants) | 72 | 73
participants | 41 | 31

3. Secondary Outcome: Objective Response Rate
Description: Best objective response of the participants from an average of 46.7 months, defined as complete or partial response according to RECIST criteria
Time Frame: 46.7 months
Measure: Number; unit: participants
Arm/Group | ZD6474 | PLACEBO
Number analyzed (Participants) | 72 | 73
participants | 6 | 4

4. Secondary Outcome: Time to Death
Description: Interim analysis time to date of randomization to date of death (data not mature at the time of this analysis, so number of deaths displayed instead.
Time Frame: time from randomization to date of death
Population: For the efficacy part, 72 were randomized to received ZD6474 and 73 placebo. For the safety part, 73 patients received at least one dose of ZD6474 and 72 placebo
Measure: Number; unit: participants
Arm/Group | ZD6474 | PLACEBO
Number analyzed (Participants) | 72 | 73
participants | 19 | 21

ADVERSE EVENTS:
Time Frame: From randomization until the end of the study, approximately up to 14 years
Description: Analysis was performed for the safety population. For participants who continued Vandetanib after the LPLV because they still benefited from it per the investigator's judgment, SAEs were collected as long as they received treatment. No non-serious adverse events were collected after LPLV for the open-label period of the study.
Groups:
- Randomized Treatment Period: Vandetanib (ZD6474): Participants received vandetanib (ZD6474) 300 mg orally once daily, until disease progression or until 12 months of stable disease during randomized treatment period, or until the end of the trial whichever comes first.
- Randomized Treatment Period: Placebo: Participants received placebo matching to vandetanib (ZD6474) tablet orally once daily, until disease progression or until 12 months of stable disease during randomized treatment period, or until the end of the trial whichever occurred first.
- Open-Label Treatment Period: Vandetanib/Vandetinib (ZD6474): Participants still receiving vandetanib (ZD6474) treatment at the end of the trial were offered the opportunity to enter the open label phase and continue to receive vandetanib (ZD6474) treatment as long as they still benefitted of it per investigator judgment or until subsequent anti-cancer therapy.
- Open-Label Treatment Period: Placebo/Vandetinib (ZD6474): Participants who experienced disease progression during the randomized phase were offered to enter the open-label phase and receive vandetanib (ZD6474) if, as long as they benefitted of it or until subsequent anti-cancer therapy.
Arm/Group | Randomized Treatment Period: Vandetanib (ZD6474) | Randomized Treatment Period: Placebo | Open-Label Treatment Period: Vandetanib/Vandetinib (ZD6474) | Open-Label Treatment Period: Placebo/Vandetinib (ZD6474)
Serious Adverse Events (participants affected / at risk) | 20/73 | 12/72 | 12/29 | 17/58
Other Adverse Events (participants affected / at risk) | 72/73 | 65/72 | 17/29 | 54/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Randomized Treatment Period: Vandetanib (ZD6474) (N=73) | Randomized Treatment Period: Placebo (N=72) | Open-Label Treatment Period: Vandetanib/Vandetinib (ZD6474) (N=29) | Open-Label Treatment Period: Placebo/Vandetinib (ZD6474) (N=58)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Angina Pectoris (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Atrioventricular Block (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bradyarrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinus Bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Torsade De Pointes (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ventricular Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Inguinal Hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intestinal Obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis Acute (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rectal Haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
General Physical Health Deterioration (General disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (2)
Bile Duct Obstruction (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis Acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gallbladder Rupture (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Drug Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchopneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Catheter Related Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dengue Fever (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 1 (1) | 1 (1) | 3 (3)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary Tract Infection Viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Drug Exposure During Pregnancy (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Femur Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Humerus Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spinal Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tibia Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Activated Partial Thromboplastin Time Prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Electrocardiogram Qt Prolonged (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tumour Lysis Syndrome (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Flank Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Groin Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Gastric Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myelodysplastic Syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tumour Haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebral Haemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebral Infarction (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cluster Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Convulsion (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysarthria (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ischaemic Stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Loss Of Consciousness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Monoparesis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spinal Cord Compression (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Transient Ischaemic Attack (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Calculus Urinary (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal Failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Interstitial Lung Disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lung Disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pleuritic Pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Cutaneous Lupus Erythematosus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Photosensitivity Reaction (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin Haemorrhage (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Randomized Treatment Period: Vandetanib (ZD6474) (N=73) | Randomized Treatment Period: Placebo (N=72) | Open-Label Treatment Period: Vandetanib/Vandetinib (ZD6474) (N=29) | Open-Label Treatment Period: Placebo/Vandetinib (ZD6474) (N=58)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 4 (5) | 1 (1) | 2 (2)
Leukopenia (Blood and lymphatic system disorders) | 4 (4) | 0 (0) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 4 (5) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 9 (12) | 7 (7) | 1 (1) | 3 (3)
Conjunctivitis (Eye disorders) | 4 (4) | 1 (1) | 0 (0) | 2 (2)
Vision Blurred (Eye disorders) | 5 (5) | 0 (0) | 0 (0) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 9 (10) | 5 (6) | 0 (0) | 6 (6)
Abdominal Pain Upper (Gastrointestinal disorders) | 1 (1) | 4 (4) | 0 (0) | 2 (3)
Cheilitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Constipation (Gastrointestinal disorders) | 5 (5) | 6 (6) | 4 (4) | 5 (5)
Diarrhoea (Gastrointestinal disorders) | 53 (66) | 12 (14) | 5 (6) | 40 (41)
Dry Mouth (Gastrointestinal disorders) | 5 (5) | 2 (2) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 4 (4) | 2 (2) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 18 (21) | 11 (11) | 1 (1) | 11 (12)
Vomiting (Gastrointestinal disorders) | 6 (7) | 5 (5) | 0 (0) | 4 (4)
Asthenia (General disorders) | 19 (19) | 16 (21) | 2 (2) | 10 (12)
Chest Pain (General disorders) | 4 (4) | 4 (4) | 0 (0) | 4 (4)
Fatigue (General disorders) | 17 (19) | 13 (13) | 3 (3) | 9 (9)
Bronchitis (Infections and infestations) | 4 (4) | 5 (6) | 1 (1) | 2 (2)
Folliculitis (Infections and infestations) | 7 (9) | 3 (3) | 1 (1) | 5 (5)
Nasopharyngitis (Infections and infestations) | 1 (1) | 4 (4) | 0 (0) | 0 (0)
Alanine Aminotransferase Increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 5 (5)
Electrocardiogram Qt Prolonged (Investigations) | 16 (17) | 0 (0) | 2 (2) | 5 (5)
Weight Decreased (Investigations) | 13 (13) | 5 (5) | 1 (1) | 6 (6)
Decreased Appetite (Metabolism and nutrition disorders) | 19 (20) | 10 (11) | 2 (2) | 9 (9)
Hypocalcaemia (Metabolism and nutrition disorders) | 6 (7) | 4 (4) | 1 (1) | 6 (6)
Hypokalaemia (Metabolism and nutrition disorders) | 9 (11) | 3 (4) | 0 (0) | 2 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 2 (2) | 2 (2)
Back Pain (Musculoskeletal and connective tissue disorders) | 4 (5) | 6 (7) | 0 (0) | 1 (1)
Bone Pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2) | 0 (0) | 3 (3)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 1 (1) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4) | 0 (0) | 1 (1)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 6 (6) | 5 (5) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 12 (13) | 14 (14) | 2 (2) | 4 (4)
Anxiety (Psychiatric disorders) | 5 (5) | 0 (0) | 1 (1) | 4 (4)
Depression (Psychiatric disorders) | 8 (8) | 0 (0) | 1 (1) | 1 (1)
Insomnia (Psychiatric disorders) | 8 (8) | 3 (3) | 0 (0) | 5 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 9 (9) | 2 (2) | 7 (7)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2) | 1 (1) | 5 (6)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 9 (11) | 2 (2) | 2 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 0 (0) | 1 (1) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 0 (0) | 3 (3)
Acne (Skin and subcutaneous tissue disorders) | 20 (21) | 6 (10) | 1 (1) | 14 (15)
Alopecia (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0) | 1 (1) | 3 (3)
Dermatitis Acneiform (Skin and subcutaneous tissue disorders) | 6 (6) | 0 (0) | 0 (0) | 2 (2)
Dry Skin (Skin and subcutaneous tissue disorders) | 12 (12) | 4 (4) | 0 (0) | 3 (3)
Eczema (Skin and subcutaneous tissue disorders) | 4 (5) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 5 (9) | 4 (4) | 1 (1) | 4 (4)
Photosensitivity Reaction (Skin and subcutaneous tissue disorders) | 13 (16) | 2 (2) | 1 (1) | 3 (3)
Pigmentation Disorder (Skin and subcutaneous tissue disorders) | 6 (8) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (4) | 4 (4) | 0 (0) | 6 (7)
Rash (Skin and subcutaneous tissue disorders) | 17 (17) | 3 (3) | 0 (0) | 11 (11)
Skin Disorder (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 2 (2) | 1 (1)
Skin Lesion (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0) | 0 (0) | 4 (5)
Hypertension (Vascular disorders) | 25 (26) | 4 (4) | 1 (1) | 19 (19)
Peripheral Coldness (Vascular disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.